CLINICAL TRIAL: NCT00347113
Title: The Effect of Schistosome and Soil-transmitted Helminth Infections on Malaria,Infection, Morbidity and Antibody Response Among School and Pre-school Children in Mwanza, Tanzania
Brief Title: Schistosome and Intestinal Worm Infections and Malaria Morbidity Among School and Pre-school Children in, Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DBL -Institute for Health Research and Development (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TAN.5.2.SAF
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2011-01

CONDITIONS: Anaemia; Malaria; Hepatosplenomegaly
Keywords: P. falciparum; malaria; schistosome infections; soil-transmitted helminths infection; anaemia; immune response; Tanzania
MeSH Terms: conditions — Anemia; Malaria | interventions — Albendazole; Praziquantel

INTERVENTIONS:
Drug: Albendazole and praziquantel

SUMMARY:
The proposed study has as the main objective to investigate the effect of schistosome and STH infections and the effect of an anthelminthic intervention on P. falciparum malaria, related anaemia and malaria antibody responses among school and pre-school children in Mwanza, Tanzania. The study will include a cross-sectional baseline survey followed by an anthelminthic intervention trial of two years duration. At baseline, prevalence and intensity of malaria, schistosome and STH infections and the prevalence of anaemia will be determined by examination of blood, faecal and urine samples. Spleen and liver size and consistency will be determined by palpation. P. falciparum specific antibodies will be determined by ELISA. All children will be treated with a single dose of praziquantel 40mg/kg and albendazole 400mg. Children selected to participate in the intervention trial will be randomized into two groups, an intervention group of 258 children which will be followed up with albendazole 400mg and praziquantel 40mg/kg at three months interval and a control group of 258 children which will be followed up with praziquantel 40mg/kg and albendazole 400mg once a year in accordance with the National Schistosomiasis and Soil-transmitted Helminths Control Programme. At 12 months and 24 months follow-up, all examinations conducted at baseline survey will be repeated.

DETAILED DESCRIPTION:
alaria is a major public health problem in tropical and subtropical countries particularly sub-Saharan Africa. Studies have shown that in Tanzania malaria, schistosome and soil-transmitted helminth infections (STH) (Hookworms, Ascaris lumbricoides and Trichuris trichiura) are co-endemic and that they share the human hosts. It has been hypothesized that co-infection with schistosomes and STH may modulate the immune response to Plasmodium falciparum leading to increased susceptibility to clinical malaria and severity of cases. The proposed study has as the main objective to investigate the effect of schistosome and STH infections and the effect of an anthelminthic intervention on P. falciparum malaria, related anaemia and malaria antibody responses among school and pre-school children in Mwanza, Tanzania. The study will include a cross-sectional baseline survey followed by an anthelminthic intervention trial of two years duration. At baseline, prevalence and intensity of malaria, schistosome and STH infections and the prevalence of anaemia will be determined by examination of blood, faecal and urine samples. Spleen and liver size and consistency will be determined by palpation. P. falciparum specific antibodies will be determined by ELISA. All children will be treated with a single dose of praziquantel 40mg/kg and albendazole 400mg. Children selected to participate in the intervention trial will be randomized into two groups, an intervention group of 258 children which will be followed up with albendazole 400mg and praziquantel 40mg/kg at three months interval and a control group of 258 children which will be followed up with praziquantel 40mg/kg and albendazole 400mg once a year in accordance with the National Schistosomiasis and Soil-transmitted Helminths Control Programme. At 12 months and 24 months follow-up, all examinations conducted at baseline survey will be repeated. If an effect of schistosome and STH infections on malaria infection and morbidity is demonstrated, control of these diseases could provide another feasible and affordable way of reducing malaria morbidity. Results of the proposed study will contribute to the understanding of the epidemiology and control of malaria in the context of other co-endemic diseases and may be important in the planning of integrated disease control strategies.

Keywords: P. falciparum, malaria, schistosome infections, soil-transmitted helminths infection, anaemia, immune response, Tanzania

ELIGIBILITY:
Inclusion Criteria:

- preschool children (>5 years of age) school children standard I-V (>7 years of age

Exclusion Criteria:

- Children with severe malaria or anaemia Children who have receuived anthelmintic treatment (< 6 months ago)

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 620 (Estimated)
Dates: Start 2006-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
incidence of malaria cases
Spleen and liver size
Hæmoglobin
P. falciparum specific antibodies (IgG3)
Prevalence and intensity of schistosome anfd intestinal helminth infections

CONTACTS AND LOCATIONS:
Overall Officials: Safari M Kinung'hi, Msc, Principal Investigator — National Insitute for Medical Research, Mwanza, Tanzania
Locations (1):
- Mwanza Medical Research Centre, Mwanza, Mwanza Region, Tanzania